CLINICAL TRIAL: NCT03762720
Title: Treatment of Muscle Injuries With Physium Therapy.
Acronym: Physium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Manuel Rodriguez Huguet, Clinical Professor, University of Cadiz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Muscle injuries
Record Dates: First submitted 2018-12-02; First posted 2018-12-04 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Injuries; Muscle, Nontraumatic
Keywords: Manual Therapy; Massage; physium; pain; range of motion; quality of life; muscle injuries
MeSH Terms: conditions — Wounds and Injuries; Pain

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CLINICAL TRIAL WITH BLIND EVALUATION BY THIRD PARTIES, LONGITUDINAL AND PROSPECTIVE.
Masking Description: Blind researcher
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physium treatment (Experimental): Patients will receive five sessions of physium therapy at 80 millibars in 30 minutes for a month
  Interventions: Device: Physium treatment

INTERVENTIONS:
Device: Physium treatment — patients will receive five sessions of physium therapy at 80 millibars in 30 minutes for one month in muscle injury and diagnosed by ultrasound and Shear Wave Elastography.

SUMMARY:
Muscle injuries are currently particularly frequent among people who participate in sports.

The diagnosis is easily made with an ultrasound study and Shear Wave Elastography.

DETAILED DESCRIPTION:
Patients of the experimental group, after diagnosis by ultrasound and Shear Wave Elastography , will receive five sessions of physium therapy at 80 millibars during one month.

The measurements of the variables visual analog scale, joint mobility through the double inclinometer device, elasticity and tissue vascularization through the ultrasound, quality of life through SF-12 questionnaire and pressure algometry will be made before, after, month and three months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged between 20 and 60 years, in an active state of pain and diagnosed with muscle breakdown.

Exclusion Criteria:

* Patients who are pregnant, have pacemakers and surgically operated in the area to be treated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2019-08-15 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Time necessary to return to full sport participation. | Baseline
  Time necessary to return to full sport participation.

SECONDARY OUTCOMES:
Time necessary to return to full sport participation. | Four weeks.
  Time necessary to return to full sport participation.
Range of motion. | Baseline and four weeks
  Measured by goniometer.
The intensity of pain | Baseline and four weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of pain, and the worst and lowest level of pain experienced in the preceding week in the area.
Pressure pain thresholds in cervical trigger points | Baseline and four weeks
  Pressure pain thresholds (PPTs) will be measured with a pressure algometer
Questionnaire SF 12 | Baseline and four weeks
  The multidimensional health related quality of life
the extent of sports-related muscle injuries | Baseline and four weeks
  Imaging is crucial to confirm and assess the extent of sports-related muscle injuries and may help to guide management.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Rodriguez Huguet, Physiotherapy, Principal Investigator — University of Cadiz

REFERENCES:
- [Background] Askling CM, Tengvar M, Thorstensson A. Acute hamstring injuries in Swedish elite football: a prospective randomised controlled clinical trial comparing two rehabilitation protocols. Br J Sports Med. 2013 Oct;47(15):953-9. doi: 10.1136/bjsports-2013-092165. Epub 2013 Mar 27. PMID 23536466
- [Background] Guermazi A, Roemer FW, Robinson P, Tol JL, Regatte RR, Crema MD. Imaging of Muscle Injuries in Sports Medicine: Sports Imaging Series. Radiology. 2017 Dec;285(3):1063. doi: 10.1148/radiol.2017174038. No abstract available. PMID 29155622
- [Background] Lee JC, Mitchell AW, Healy JC. Imaging of muscle injury in the elite athlete. Br J Radiol. 2012 Aug;85(1016):1173-85. doi: 10.1259/bjr/84622172. Epub 2012 Apr 11. PMID 22496067
- [Background] Sporea I, Lie I. Shear wave elastography. Ultraschall Med. 2012 Aug;33(4):393-4. No abstract available. PMID 23045734
- [Background] Kinser AM, Sands WA, Stone MH. Reliability and validity of a pressure algometer. J Strength Cond Res. 2009 Jan;23(1):312-4. doi: 10.1519/jsc.0b013e31818f051c. PMID 19130648
- [Background] Bonilla D, Hortalá G, Temporal D, CarréLlopis C. PHYSIUM in thetreatment of pain in patientswithchroniclow back pain. FisioGlía. 2015;2(3):50-55.
- [Background] Maquet D, Croisier JL, Demoulin C, Crielaard JM. Pressure pain thresholds of tender point sites in patients with fibromyalgia and in healthy controls. Eur J Pain. 2004 Apr;8(2):111-7. doi: 10.1016/S1090-3801(03)00082-X. PMID 14987620
- [Background] Ko SJ, Kim H, Kim SK, Park K, Lee J, Lee BJ, Oh J, Lee K, Park JW. Reliability and Validity of Modified Algometer in Abdominal Examination. Evid Based Complement Alternat Med. 2016;2016:3052954. doi: 10.1155/2016/3052954. Epub 2016 Mar 17. PMID 27073401
- [Background] Chesterton LS, Barlas P, Foster NE, Baxter DG, Wright CC. Gender differences in pressure pain threshold in healthy humans. Pain. 2003 Feb;101(3):259-266. doi: 10.1016/S0304-3959(02)00330-5. PMID 12583868
- [Background] Vilagut G, Valderas JM, Ferrer M, Garin O, Lopez-Garcia E, Alonso J. [Interpretation of SF-36 and SF-12 questionnaires in Spain: physical and mental components]. Med Clin (Barc). 2008 May 24;130(19):726-35. doi: 10.1157/13121076. Spanish. PMID 18570798
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Ayala F, De Ste Croix M, Sainz de Baranda P, Santonja F. Acute effects of static and dynamic stretching on hamstrings' response times. J Sports Sci. 2014;32(9):817-25. doi: 10.1080/02640414.2013.861606. Epub 2014 Jan 10. PMID 24405028
- [Background] Ohno Y, Fujimoto T, Shibata Y. A New Era in Diagnostic Ultrasound, Superb Microvascular Imaging: Preliminary Results in Pediatric Hepato-Gastrointestinal Disorders. Eur J Pediatr Surg. 2017 Feb;27(1):20-25. doi: 10.1055/s-0036-1593381. Epub 2016 Oct 3. PMID 27699732